CLINICAL TRIAL: NCT00056420
Title: Spatiotemporal Dynamics of Cortical Connectivity Involved in Tics and Voluntary Movements in Patients With Tourette's Syndrome and Chronic Motor Tic Disorder: An EEG Study
Brief Title: Brain Dynamics Involved in Generating Tics and Controlling Voluntary Movement
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030126; 03-N-0126
Record Dates: First submitted 2003-03-12; First posted 2003-03-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-01-22

CONDITIONS: Tourette Syndrome; Tic Disorders
Keywords: Tourette's Syndrome; Tic Disorder; (EEG) Electroencephalography; Event-Related Desynchronization/Synchronization; Coherence; Tourette's; Tourette Syndrome; Healthy Volunteer; HV
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders

SUMMARY:
This study will use electroencephalography (EEG) and electromyography (EMG) to examine how the brain generates tics and controls voluntary movement in patients with Tourette's syndrome and chronic motor tic disorder. EEG records the electrical activity of the brain. For this test, a cap with built-in electrodes is placed on the subject's head, and the electrodes are connected to a monitor that records the brain activity. EMG records muscle activity using electrodes placed on the skin over muscles on the fingers or above the outer corner of the eyes.

Healthy normal volunteers and patients with Tourette's syndrome and chronic motor tic disorder between 21 and 65 years of age may be eligible for this 2- to 3-hour study. Each candidate will be screened with a medical history, physical and neurological examinations, and a questionnaire that screens for psychiatric disorders.

During EEG and EMG recordings, participants undergo the following tasks while seated comfortably in a sound-shielded room:

Patients

* Finger task: Patients raise their index finger once every 10 seconds for about 25 minutes.
* Tic evaluation and mimicking: Patients allow their tics to occur as they do naturally. After each tic, they report whether the tic was voluntary and whether it was preceded by a sensation of urge. They then mimic tics that they normally have, at a rate of about once every 10 seconds.
* Tic suppression task: Patients suppress tics they normally have for several minutes. They then allow the tics to occur naturally, without attempting to suppress them.

Normal Volunteers

* Finger task: Volunteers raise their index finger once every 10 seconds for about 25 minutes.
* Open eye task: Volunteers keep their eyes open for a minute or so, and then resume blinking as often as feels comfortable. The process is repeated several times.

DETAILED DESCRIPTION:
This study examines the spatiotemporal dynamics of cortical functional interconnectivity involved tics and voluntary movement in patients with Tourette's syndrome or chronic motor tic disorder. By employing a combination of EEG methods that utilize analyses in the domains of both frequency (e.g., event-related desynchronization/synchronization (ERD/ERS), event-related partial coherence, phase coherence) and time (e.g., event-related partial correlation), we intend to determine

1. Whether the cortical neurocircuitry involved in the performance of a simple, voluntary motor task differs in patients with tic disorders from that of healthy volunteers;
2. Whether the network involved in the generation of unwanted tics differs from that of normal voluntary movement (i.e., mimicked tics); and
3. What role, if any, premonitory urge and/or tic suppression plays in the modulation of this neurocircuitry.

ELIGIBILITY:
* INCLUSION CRITERIA:

HEALTHY VOLUNTEERS:

Healthy volunteers are between the ages of 21 and 65 years.

PATIENTS:

Patients will have clinically documented Tourette's syndrome or chronic motor tic disorder as defined by DSM-IV-TR and evaluation of tic severity using the Yale Tic Scale. This criterion will be established by preliminary screening in the NINDS Movement Disorders Outpatient Clinic. Regarding co-morbid disorders such as ADHD and OCD, we will accept a mild degree of ADHD and mild to moderate degree of OCD. These disorders will be established by a psychiatrist using below listed scales and criteria.

Structure Clinical Interview for (DSMIV SCID) will be administered to all subjects to ensure that strict DSM-IV criteria for Tourette Syndrome have been met and to assess for possible comorbid psychiatric disorders.

Given the high rate of comorbidity of Obsessive Compulsive Disorder (OCD) and Attention Deficit/Hyperactivity Disorder (ADHD) in Tourette's syndrome, it may not be possible to exclude persons with these disorders. Hence, only those with no more than mild to moderate severity of symptoms will be accepted into the study. This will be ascertained using the following instruments and their respective cut-off scores:

Y-BOCS (Goodman et al, 1989) a 10 item scale with a range of 0 - 4 and maximum possible score of 40 (0-7: subclinical; 8 - 15: mild; 16 -23: moderate; 24 - 31 severe; 32 - 40: extreme). Inclusion criteria: 23 or below.

ADHD Behavior Checklist for Adults (Barkley, 1995, Murphy and Barkley, 1995): An 18 Item checklist with 9 Inattention items and 9 Hyperactive/impulsive items ranging 0 - 3 (0: never or rarely 1: sometimes 2: often and 3: very often ). Items answered often or very often are scored as present. With age, the threshold criterion for presence of ADHD become lower and is currently accepted as follows:

Age Range; Inattention Items; Hyperactive and Impulsive Items respectively:

21-29 years; 4 of 9; 5 of 9

30-49; 4 of 9; 4 of 9

50 and over; 3 of 9; 3 of 9

Inclusion Criteria:

Age Range; Inattention Items; Hyperactive and Impulsive Items respectively:

21-29 years; 3 or below; 4 or below

30-49; 3 or below; 3 or below

50 and over; 2 or below; 2 or below

EXCLUSION CRITERIA IN HEALTHY VOLUNTEERS AND PATIENTS:

The following subjects will be excluded from the study:

1. Subjects younger than 21 or older than 65 years, as EEG studies have shown findings to vary with neurodevelopment and age.
2. Subjects with 1) major depression, 2) bipolar disorder, or 3) psychotic disorder. Such coexisting neuropsychiatric disorders may lead to unnecessary confounds of the data.
3. Subjects taking benzodiazepines, anti-depressant or neuroleptic medications (such medications are known to affect EEG and may thus confound data)
4. Subjects with major acute or chronic illness (experimental setting may be unnecessarily uncomfortable or unpleasant)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54
Dates: Start 2003-03-10; Study Completion 2009-01-22

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Biswal B, Ulmer JL, Krippendorf RL, Harsch HH, Daniels DL, Hyde JS, Haughton VM. Abnormal cerebral activation associated with a motor task in Tourette syndrome. AJNR Am J Neuroradiol. 1998 Sep;19(8):1509-12. PMID 9763386
- [Background] Braun AR, Stoetter B, Randolph C, Hsiao JK, Vladar K, Gernert J, Carson RE, Herscovitch P, Chase TN. The functional neuroanatomy of Tourette's syndrome: an FDG-PET study. I. Regional changes in cerebral glucose metabolism differentiating patients and controls. Neuropsychopharmacology. 1993 Dec;9(4):277-91. doi: 10.1038/npp.1993.64. PMID 8305128
- [Background] Brown P, Marsden CD. What do the basal ganglia do? Lancet. 1998 Jun 13;351(9118):1801-4. doi: 10.1016/s0140-6736(97)11225-9. PMID 9635969